CLINICAL TRIAL: NCT01361243
Title: NOURISHing Families to Promote Healthy Eating and Exercise in Overweight Children
Brief Title: NOURISH+: Nourishing Our Understanding of Role Modeling to Improve Support and Health
Acronym: NOURISH+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM13468; R01HD066216-01A1 (NIH)
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Overweight and Obesity
Keywords: Pediatric Overweight; Pediatric Obesity
MeSH Terms: conditions — Overweight; Obesity; Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NOURISH+ (Experimental): Participants will receive a 6-week face-to-face intervention, NOURISH+. Weekly topics teach parents skills to role model and encourage healthy lifestyle behaviors for their children.
  Interventions: Behavioral: NOURISH+
- Wellness Group (Placebo Comparator): Participants will receive an in-person "Family Wellness Night" followed by 6 mailings of information regarding pediatric overweight and obesity.
  Interventions: Behavioral: Wellness Group

INTERVENTIONS:
Behavioral: NOURISH+ — 6 week face-to-face parent intervention.
  Arms: NOURISH+
Behavioral: Wellness Group — 1 week face-to-face family group followed by 6 informational mailings on childhood overweight and obesity.
  Arms: Wellness Group

SUMMARY:
The purpose of this study is to evaluate the efficacy of a parent intervention (NOURISH+) aimed at reducing the problem of overweight and obesity in children.

DETAILED DESCRIPTION:
Pediatric overweight is a national public health concern. The percentage of overweight children in the U.S. between the ages of 5 and 11 has nearly tripled in the last 3 decades. African American children are particularly at risk. Pediatric overweight is associated with numerous physical and psychological health problems. Moreover, overweight children are at significant risk for obesity in adulthood. Thus, a focus on pediatric overweight is an important step in the prevention of adult obesity.

Despite the urgent need for pediatric overweight interventions, outcomes of some of the most rigorous treatments are, at best, mixed. Although research has found that including parents in interventions for pediatric overweight has positive effects on outcomes, parental involvement is usually limited. Moreover, relatively few studies have included sufficient numbers of lower-SES, African American participants, a group at increased risk for pediatric overweight and associated complications. This study will evaluate the efficacy of an intensive intervention targeting ethnically diverse parents of overweight, children ages 5-11 (NOURISH-Nourishing Our Understanding of Role Modeling to Improve Support and Health).

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregivers must be at least 18 years old
* Parents/caregivers must have a child between the ages of 5 and 11 with a BMI > the 85th percentile, who primarily resides in the caregiver's home
* Parents/caregivers need to speak English, be able to follow basic instructions, and perform simple exercises

Exclusion Criteria:

* Non-ambulatory parents/caregivers
* Pregnant parents/caregivers
* Parents/caregivers who have a medical condition that might be negatively impacted by exercise
* Parents/caregivers who have a psychiatric diagnosis that would impair their ability to respond to assessments or participate in a group
* Parents whose children have a medical or developmental condition that precludes weight loss using conventional diet and exercise methods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2011-04; Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Child BMI | baseline, post-testing, 4-month, and 10-month follow-up

SECONDARY OUTCOMES:
Child dietary intake, quality of life, and physical activity | baseline, post-testing, 4-month, and 10-month follow-up
Parental BMI, dietary intake, and physical activity levels | baseline, post-testing, 4-month, and 10-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne E Mazzeo, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwitowski M, Bean MK, Mazzeo SE. An exploration of factors influencing attrition from a pediatric weight management intervention. Obes Res Clin Pract. 2017 Mar-Apr;11(2):233-240. doi: 10.1016/j.orcp.2016.08.002. Epub 2016 Aug 17. PMID 27544283